CLINICAL TRIAL: NCT05463874
Title: Teaching Adolescents with Type 1 Diabetes Self-compassion to Reduce Diabetes Distress: a Randomized Controlled Trial
Brief Title: Teaching Adolescents with Type 1 Diabetes Self-compassion
Acronym: TADS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); Brain Canada (Other)
Responsible Party: Principal Investigator, Marie-Eve Robinson, Principal Investigator, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22/08E
Record Dates: First submitted 2022-07-12; First posted 2022-07-19 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mindful Self-Compassion Arm (Experimental): Participants in this arm will participate in an 8-week virtual mindful self-compassion program.
  Interventions: Behavioral: Mindful Self-Compassion Program
- Wait-list Control Arm (No Intervention): Participants in this arm will receive usual clinical care and will have the opportunity to participate in the mindful self-compassion program at the end of the study.

INTERVENTIONS:
Behavioral: Mindful Self-Compassion Program — The intervention consists of 8 sessions, one per week for 8 weeks, that last 1 hour and 30 minutes each. These sessions will cover a variety of mindfulness and self-compassion practices, such as dealing with difficult emotions and developing a kind inner voice.
  Arms: Mindful Self-Compassion Arm

SUMMARY:
The purpose of this study is to see if a mindful self-compassion program given virtually can improve emotional distress for youth with type 1 diabetes, compared to routine care as usual.

DETAILED DESCRIPTION:
Background: Type 1 diabetes (T1D) is a chronic, life-long condition. Youth with T1D must monitor their blood sugar levels, nutrition, physical activity, and other daily activities. They also need insulin multiple times per day.

Diabetes distress can happen when all the worry, frustration, anger, and burnout make it hard for people with diabetes to take care of themselves and keep up with the daily demands of their condition. Most youth with T1D experience diabetes distress and over one third experience severe diabetes distress.

Self-compassion is a practice that involves acting the same way towards yourself as you would with friends and loved ones, and that you are kind and understanding towards yourself. Since self-compassion is a skill that can be taught, we hypothesize that it could be a strategy to improve mental health issues in youth with T1D, like diabetes distress.

Objectives: The aim of our study is to assess the effectiveness of a mindful self-compassion program on improving the diabetes distress experienced by youth aged 12-17 years with T1D. We will compare if diabetes distress 3 months after enrolment in the study is different among youth that received the mindful self-compassion program versus the ones that did not. We will also assess the effect of the program on anxiety, depression, diabetes-related disordered eating, and suicidal ideation. Finally, we will explore the effect of the program on blood sugar control, and if the effects change over time.

Methods: Our study will be a randomized controlled trial of youth aged 12-17 years, with a diagnosis of T1D. Participants will be recruited from the diabetes clinic at the Children's Hospital of Eastern Ontario (CHEO) and randomized to the mindful self-compassion program or a wait-list control group. The mindful self-compassion program will consist of weekly virtual 1.5-hour sessions/workshops for 8 weeks, led by a trained facilitator. It will cover a variety of self-compassion practices, such as dealing with difficult emotions and developing a kind inner voice. The wait-list group will be offered the mindful self-compassion program once the experimental period of the study is over.

Outcomes in both groups will be assessed at the start of the study, 8-weeks, and at 3-, 6-, and 12- months. Participants showing signs of suicidal ideation or severe depression will be assessed clinically by the study doctor and appropriate follow up actions will be taken.

ELIGIBILITY:
Inclusion Criteria:

* Between 12-17 years of age
* Diagnosed with type 1 diabetes at least 6 months prior to enrollment
* Able to provide informed consent

Exclusion Criteria:

* Unable or unwilling to provide informed consent
* Do not speak English or French with enough fluency to complete all study related tasks
* Presence of an intellectual disability that would preclude participation in the MSC intervention, as assessed by the treating physician
* Lifetime diagnosis of a serious mental illness given by a clinician (e.g., psychotic or bipolar disorders), as these often involve intensive treatments with psychological and/or pharmacologic implications, which may confound our results.
* Presence of acute suicidality at the time of enrollment (if a patient reports suicidality on the baseline questionnaires, a same-day assessment will be conducted to assess for acute suicidality. If present, the patient will receive immediate clinical attention and will no longer be eligible to participate in the study).
* Active participation in another mental health intervention trial.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 141 (Actual)
Dates: Start 2022-10-04 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Diabetes Distress as measured by the Problem Areas in Diabetes - Teen Version (PAID-T) | 3 months
  Diabetes distress as measured by the PAID-T will be compared in those who complete the MSC program to those in the wait-list control group at 3 months. Scores can range from 26-156, with scores of <70, 70-90, and >90 representing none-to-mild, moderate, and severe diabetes distress, respectively.

SECONDARY OUTCOMES:
Anxiety as measured by the Generalized Anxiety 7-item scale (GAD-7) | 3 months, 12 months
  Anxiety as measured by the GAD-7 will be compared between those who complete the MSC program and those in the wait-list control group at 3 months and at 12 months. The GAD-7 is scored from 0-21, with 0-4, 5-9, 10-14, and 15-21 indicating minimal, mild, moderate, and severe anxiety symptoms respectively.
Depression as measured by the Patient Health Questionnaire (PHQ-9) | 3 months, 12 months
  Depression as measured by the PHQ-9 in those who complete the MSC program compared to those in the wait-list control group will be assessed at 3 months and at 12 months. PHQ-9 scores range from 0-27, and in adolescents, scores of 0-4, 5-10, 11-14, 15-19, and ≥20 indicate absence of depression, mild depression, moderate depression, moderately severe depression, and severe depression respectively.
Disordered eating as measured by the Diabetes Eating Problem Survey, revised version (DEPS-R) | 3 months, 12 months
  Disordered eating as measured by the DEPS-R will be compared in those who complete the MSC program and those in the wait-list control group at 3 months and at 12 months. The DEPS-R is scored 0-80, with higher scores indicating more disordered eating behaviors and a score of ≥20 considered a positive screen for disordered eating behaviours.
Suicidal ideation as measured by the Patient Health Questionnaire (PHQ-9) | 3 months, 12 months
  Suicidal ideation in those who complete the MSC intervention will be compared to those in the wait-list control group at 3 months and at 12 months. Suicidal ideation will be assessed using one question on the PHQ-9, which asks the respondent if they have had thoughts that they would be better off dead, or of hurting themselves in the previous two weeks. This question is scored on a scale of 0 (not at all) to 3 (nearly every day). In line with previous use of the PHQ-9, we will consider any score of >0 to be indicative that suicidal ideation is present.
Diabetes distress as measured by the Problem Areas in Diabetes - Teen version (PAID-T) | 12 months
  Diabetes distress as measured by the PAID-T will be compared in those who complete the MSC program to those in the wait-list control group at 12 months. Scores can range from 26-156, with scores of <70, 70-90, and >90 representing none-to-mild, moderate, and severe diabetes distress, respectively.

OTHER OUTCOMES:
Interaction term of time and diabetes distress | Baseline, 8 weeks, 3 months, 6 months, 12 months
  We will assess whether the effect of the MSC intervention on diabetes distress, as measured by the Problem Areas In Diabetes - Teen version (PAID-T) changes over time by exploring the interaction of time (i.e., study timepoint) with diabetes distress.
Hemoglobin A1c | Baseline, 12 months
  HbA1c is a measure of the average blood glucose levels over the previous 3 months and is a routinely followed biochemical marker used to gauge metabolic control in individuals with T1D. We will explore change in HbA1c over the duration of our trial as mental health morbidity has been associated with higher HbA1c levels. A change of more than 0.5% will be considered clinically significant.
Time in Range | Baseline, 8 weeks, 3 months, 6 months, 12 months
  Time in range is a metric that denotes the proportion of time that a person's glucose level is within a desired target range. Continuous glucose monitoring (CGM) devices are required to calculate time in range. Fourteen days of data from CGM provides a good approximation of glucose data; time in range will allow us to evaluate the glucose control at the various study time points.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Eve Robinson, MD, MSc, Principal Investigator — Children's Hospital of Eastern Ontario
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontatrio, Canada

IPD SHARING:
Plan to Share IPD: No
IPD will be made available upon reasonable request from other researchers.

REFERENCES:
- [Derived] Dover S, Ahmet A, Bluth K, Feldman BM, Goldbloom EB, Goldfield GS, Hamilton S, Imran O, Khalif A, Khatchadourian K, Lawrence S, Leonard A, Liu K, Ouyang Y, Peeters C, Shah J, Spector N, Zuijdwijk C, Robinson ME. Teaching Adolescents With Type 1 Diabetes Self-Compassion (TADS) to Reduce Diabetes Distress: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2023 Dec 26;12:e53935. doi: 10.2196/53935. PMID 38048480